CLINICAL TRIAL: NCT01273636
Title: Concurrent Endometrial Cancer With Endometrial Hyperplasia or Endometrial Intraepithelial Neoplasia - Focus on Risk Factors Analysis
Brief Title: Risk Factors for Concurrent Endometrial Carcinoma in Patients With a Curettage Diagnosis of Endometrial Hyperplasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chi-An Chen/Professor, National Taiwan Unviersity Hospital
Other Study IDs: 200712018R
Record Dates: First submitted 2008-08-14; First posted 2011-01-10 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2010-12

CONDITIONS: Endometrial Carcinoma
Keywords: Endometrial hyperplasia; Hysterectomy; Endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective: To examine the risk factors for coexisting endometrial carcinoma in patients with endometrial hyperplasia.

Method: Seventy-seven patients who received hysterectomy for endometrial hyperplasia were enrolled and divided into the non-endometrial carcinoma group (57) and the endometrial carcinoma group (20) depending on the final pathology. Clinical variables were analyzed.

DETAILED DESCRIPTION:
We retrospectively reviewed the cases of seventy-seven patients who had hysterectomies for endometrial hyperplasia between January 1996 and September 2006 at the Department of Obstetrics and Gynecology, National Taiwan University Hospital. A preoperative pathologic diagnosis of endometrial hyperplasia was obtained by D&C (dilation and curettage) in all patients. Twenty of them were diagnosed as having endometrial carcinoma in their hysterectomy specimens. All of the specimens were reviewed by a gynecologic pathologist.

Depending on the final pathologic reports of hysterectomy, we divided the seventy-seven patients into two groups - the non-endometrial carcinoma group and the endometrial carcinoma group. Fifty-seven of the studied patients were in the non-endometrial carcinoma group and twenty were in the endometrial carcinoma group. As already mentioned above, we investigated them by clinical parameters including age, menopausal status, obstetrical history, medical history of diabetes and hypertension, BMI (body mass index) and preoperative pathology of D&C.

The clinical and pathologic characteristics of the twenty patients diagnosed as having endometrial carcinoma postoperatively were also reviewed. Initial manifestation, histological grading of the carcinoma, the depth of myometrial invasion, with or without adjuvant radiotherapy and recurrence were included. The histological grading of endometrial carcinoma was based on FIGO ( International Federation of Gynecology and Obstetrics ) definitions. The BMIs of the patients with endometrial carcinoma were also analyzed by the receiver operating characteristic curve. The Research and Ethics Committee of National Taiwan University Hospital approved this study.

Statistical analyses were performed with the Independent-Samples T test and the Mann-Whitney test. Subsequently, multivariate analysis of risk factors was also employed with Binary logistic regression model to obtain the adjusted odds ratio (OR) and 95% confidence interval (CI) for selective variables. P<0.05 was defined as significant.

ELIGIBILITY:
Inclusion Criteria:

* Endometrial hyperplasia patient having hysterectomy with or without bilateral salpingo-oophorectomy

Exclusion Criteria:

* none

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We retrospectively reviewed the cases of seventy-seven patients who had hysterectomies for endometrial hyperplasia between January 1996 and September 2006 at the Department of Obstetrics and Gynecology, National Taiwan University Hospital. A preoperative pathologic diagnosis of endometrial hyperplasia was obtained in all patients.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2005-01; Primary Completion 2006-01 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
The prognosis of patients diagnosed as endometrial carcinoma after hysterectomy. | From carcinoma diagnosed to the last patient follow-up or death till June, 2011

CONTACTS AND LOCATIONS:
Overall Officials: Chi An Chen, M.D., Study Chair — Department of Obstetrics and Gynecology, National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - Chi-An Chen, Taipei, Taiwan
  - Chi-An Chen, Taipei